CLINICAL TRIAL: NCT05461547
Title: Pre-Hospital Lung Ultrasound Impact on Diagnosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Awaiting grant funding to continue
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Frances Russell, Associate Professor Emergency Medicine, Indiana University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 15954
Record Dates: First submitted 2022-06-30; First posted 2022-07-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Heart Failure
Keywords: ultrasound; prehospital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Usual Care (Other)
  Interventions: Other: Usual Care
- Lung Ultrasound (Experimental)
  Interventions: Diagnostic Test: Lung Ultrasound

INTERVENTIONS:
Diagnostic Test: Lung Ultrasound — LUS will be performed and interpreted in real-time to guide acute management.
  Arms: Lung Ultrasound
Other: Usual Care — Usual care to decide diagnosis and treatment
  Arms: Usual Care

SUMMARY:
Acute heart failure (AHF) is a major reason patients seek emergency care and is a significant public health burden. The ability to differentiate AHF from other etiologies of dyspnea remains a challenge as symptoms and physical exam findings overlap, especially in the pre-hospital setting where diagnostic tools are not readily available. The inability to differentiate AHF from other causes of dyspnea leads to misdiagnosis, delays in diagnosis, and ultimately delays in appropriate treatment. Delays in initiating HF therapies is associated with poor outcomes including higher rates of in-hospital mortality and longer hospital length of stay. Optimizing treatment for AHF in the pre-hospital setting is associated with increased survival and lower rates of hospital re-admission. Thus, accurate diagnosis and early treatment for AHF in the pre-hospital setting remains a critical unmet need. Lung ultrasound (LUS), through assessment of B-lines, allows for an easy and accurate method for detection of pulmonary congestion seen in AHF patients. Although multiple studies have shown LUS is easy to learn, there is a paucity of data assessing clinical impact of LUS in the pre-hospital setting. The investigators hypothesize that the use of LUS by pre-hospital personnel will improve accuracy for detecting AHF in the pre-hospital setting when compared to usual care (no LUS).

Specific Aims: To determine if the use of pre-hospital LUS improves diagnostic accuracy for detecting AHF in patients transported by emergency medical services (EMS) for acute dyspnea when compared to usual care (no LUS).

DETAILED DESCRIPTION:
Prospective, randomized study using a phased implementation on patients being transported by EMS to the hospital for acute dyspnea. The investigators will include adults (>17yo) with a chief complaint of dyspnea and at least one of the following: bilateral lower extremity edema, orthopnea, wheezing or rales on auscultation, increased work of breathing, tachypnea (RR>20) or hypoxia (oxygen saturation <92%). Patients with fever (>100.4F), systolic blood pressure <90mmHg, those requiring immediate intubation, those found to have ST elevation myocardial infarction on EKG, or pregnant will be excluded. Eligible patients will be enrolled in the pre-hospital setting over a 12-month period. Randomization that will occur at the ambulance level using a stepped wedge cluster randomization trial design. Twenty-six full-time paramedics previously trained in LUS will perform a 2 or 4-view imaging protocol and interpret images in real-time to guide acute management. The diagnosis of AHF on LUS will be defined as bilateral B-lines (>2 B-lines in a zone in each hemi-thorax). A hospital diagnosis of AHF versus not HF will be determined through independent chart review by two blinded physicians and will serve as the criterion standard for final diagnosis. Diagnosis by paramedics, whether LUS was used, and treatment given pre-hospital will be tracked in ESO (an online EMS clinical documentation system). For the primary aim the investigators will compare pre-hospital provider diagnosis to final diagnosis to determine accuracy with and without the use of LUS.

Expected Results: The investigators anticipate the use of prehospital LUS will improve diagnostic accuracy for detecting AHF. This pilot study will set the groundwork for future larger studies assessing the clinical impact of prehospital LUS.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>17yo) with a chief complaint of shortness of breath.

Exclusion Criteria:

* We will exclude patients with hypotension (SBP <90), an EKG showing ST-segment elevation, fever >100.4F, trauma or who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of pre-hospital providers for identifying AHF versus not AHF | 3 years
  Pre-hospital providers will diagnose AHF or not HF with and without LUS. Diagnostic accuracy will be determined by comparing pre-hospital diagnosis to hospital diagnosis of AHF versus not AHF through independent chart review.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No